CLINICAL TRIAL: NCT06262646
Title: Effectiveness of Video-conferencing Focused Acceptance and Commitment Therapy Compared With Standard Parenting Advice for Parents of Young Children With Special Needs: A Randomized Clinical Trial
Brief Title: Video-conferencing FACT for Young Children With Special Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hong Kong Christian Service (Other); Hong Kong Federation of Youth Groups (Unknown); Hong Kong Young Women's Christian Association (Other); Yang Memorial Methodist Social Service (Other); Hong Kong Sheng Kung Hui Welfare Council Limited (Other)
Responsible Party: Principal Investigator, Yuen Yu CHONG, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NTEC-2023-677
Record Dates: First submitted 2024-02-01; First posted 2024-02-16 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder; Specific Learning Disorder; Communication Disorders; Motor Disorders
Keywords: Acceptance and Commitment Therapy; Children with Special Needs; Parental psychological health; Parenting stress; Psychological Interventions; Randomized controlled trial
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Specific Learning Disorder; Communication Disorders; Motor Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Two-arm Randomised Controlled Trial (RCT) with a repeated-measures parallel-group design
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Eligible parents consenting to participate will be randomly assigned to either the FACT or Control Group in a 1:1 ratio, using the permuted block size of 6 through sequentially numbered, opaque and sealed envelopes with number cards (1=intervention, 2=control). A separate set of random numbers, concealed from the research team and RAs, will be generated by a statistician. Clerical staff uninvolved in the project will administer the randomisation. The research assistant (RA-1), blinded to subject selection, will open the envelopes only after informed consent and baseline assessments are completed. The research assistant (RA-2) is also blinded to group assignments and will conduct assessments/evaluations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FACT Group (Experimental): Parents will receive 4-6 FACT consultation sessions, one weekly session, 45-60 mins per session. These sessions will be one-on-one, conducted face-to-face or via video conferencing.
  Interventions: Behavioral: Focused Acceptance and Commitment Therapy
- Control Group (Active Comparator): Parents will receive standard parenting advice about positive parenting tips recommended by the Child Assessment Services under the Department of Health.
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Focused Acceptance and Commitment Therapy — Trained FACT interventionists will be guided by manualized FACT intervention to identify how many psychopathological processes need support and which ACT process(es) need to work on first, then offer parents process-matched ACT intervention strategies following the principles of FACT. The intervention strategies include ACT metaphors, experiential exercises, audio-guided mindfulness exercises, guided imagery exercises and value clarification exercises. The FACT steps in each session depend on the client's situation/stage.
  Other Names: FACT
  Arms: FACT Group
Other: Control Group — Both study groups will receive standard family support from collaborating NGOs.
  Arms: Control Group

SUMMARY:
Objective: This RCT evaluates the efficacy of Focused Acceptance and Commitment Therapy (FACT) delivered via videoconferencing for parents of special needs children, targeting reducing parental stress (primary outcome), symptoms of depression and anxiety, as well as psychological flexibility.

Background: Parental caregiving for children with special needs is associated with significant stress, potentially impairing parental and familial functioning. Acceptance and Commitment Therapy (ACT) has shown promise in bolstering mental health across diverse populations. Preliminary findings from a feasibility trial (NCT05803252) suggest the potential of FACT in this context.

Methods: Expanding upon prior research, this definitive RCT compares FACT to standard parenting advice, correcting for earlier limitations through increased sample size and rigorous methodology. Assessments will be conducted at baseline, post-intervention (4-8 weeks), and 6-month follow-up.

Results: The study anticipates that FACT will demonstrate superior outcomes in promoting well-being among parents compared to parenting advice alone.

Conclusion: By leveraging videoconferencing for therapy delivery, the RCT aims to improve access to mental health interventions and emphasize the importance of psychological health among parents of special needs children. This could foster greater recognition and proactive management of mental health within this population.

DETAILED DESCRIPTION:
INTRODUCTION Children with special health care needs (SHCN) are defined as those who have/are at high risk for having chronic physical, developmental, behavioural, and/or emotional conditions requiring specialized and considerable health and related services of type(s)/amount beyond 12 months. Although there is no central registry for children with SHCN in Hong Kong, for pre-schoolers with developmental conditions, there has been a prevailing rate of newly diagnosed cases of special health care needs children in Hong Kong (17,193 in 2019) and an annual increase rate of 6.2-10.7% in the number of referred cases for speciality follow-up services in the Child Assessment Centre under the Department of Health.

Parents of children with special health care needs (SHCN) have always been under tremendous pressure to take care of their children. They have been experiencing significant caregiving difficulties, such as scheduling and accompanying multiple follow-ups for rehabilitation and functional recovery and managing a child's symptoms and problematic behaviours. In addition, parenting stress has been known to affect parent-child interactions, increase negative parenting behaviours such as harsh, permissive, or neglectful parenting, and impair the parent's capacity to respond to the demands of the child's illness, which may, in turn, exacerbate the child's health problem and well-being. The above shows an emerging need to provide and expand mental health care support to these parents and children in a format that is sustainable and undisrupted by the restriction measures caused by the pandemic.

In literature, there has been increasing evidence supporting the efficacy of Acceptance and Commitment Therapy (ACT) on mental health in different population groups, including healthy individuals, parents, children, and those with mental health problems. Though the result was promising, the previous clinical trials in Hong Kong showed a limited effect size. This is due to the need for extensive manpower in ACT intervention, yet there are very limited trained ACT interventionists in Hong Kong. On top of that, past interventions have failed to target impaired psychopathological processes as well as identify and determine which psychopathological processes require intervention in the first place. This study aims to overcome the limitations mentioned above.

BACKGROUND Acceptance and Commitment Therapy Acceptance and Commitment Therapy (ACT) is a new form of mindfulness- and values-based behavioural therapy. In literature, ACT has demonstrated proven efficacy on the mental health symptoms of people diagnosed with depression and anxiety, as well as parents of children with developmental conditions (e.g., autism spectrum disorders and developmental delays).

The PI and her research team have conducted the first ACT clinical trial for Hong Kong parents of children with asthma, showing that a 4-session parental training programme using group-based ACT integrated with asthma education was more effective than education alone for improving parental psychological well-being, parental asthma management self-efficacy and childhood asthma morbidity. Currently, the PI's team is actively expanding the research studies in ACT to other population groups in Hong Kong, such as parents and their children with asthma comorbid with ADHD, parents of children with autism spectrum disorder, parents and their children with eczema and patients with early psychosis. In addition, our team has extensive experience in conducting clinical trials using mindfulness-based interventions for family caregivers and/or individuals with schizophrenia and dementia, as well as evaluating the efficacy of self-help programmes for facilitating patients with recent-onset psychosis to acquire better problem-solving abilities.

The results mentioned above encouraged the development of ACT in the service of parents in Hong Kong. Yet previous studies show that ACT could be a long-term intervention and require frequent follow-up, which would increase the burden on healthcare professionals. A recent systematic review of ACT for clients with anxiety and depression has highlighted the issues of multiple sessions (at least 6-8 weekly sessions for a completed treatment for one client) and notable attrition (with a mean of 19.2%, ranging from 0-60.8%). This could be attributed to the lack of targeting at parents' psychological needs by assessing how many psychopathological processes parents require for support and what process(es) they need to work on first. Given Hong Kong's development, there are exceptionally few trained ACT interventionists, and the time-consuming intervention would not be feasible.

The proposed study aims to overcome the above limitation by adopting Focused Acceptance and Commitment Therapy (FACT), which is a time-limited and brief intervention that provides systematic ACT intervention targeting parents' psychological needs and offering customized processed-matched ACT intervention.

Focused Acceptance and Commitment Therapy (FACT) FACT is a new model of brief therapy that is a highly condensed version of Acceptance and Commitment Therapy. As suggested by Strosahl, Robinson and Gustavsson, FACT aims to orient clients to observe and accept distressing experiences and unwanted emotions rather than attempting to suppress and control them, helping clients identify and connect with personal values and engaging in taking committed actions that are consistent with clients' own values through increasing one's psychological flexibility. In clinical trials, it was shown that brief ACT interventions were able to produce long-term results. A review of forty ACT components studies done by Levin, Hildebrant, Lillis & Hayes showed an average weighted effect size of d= 0.70. The effect size of the brief intervention laid the way for the development of FACT. A study done by Strosahl, Hayes, Bergan, & Romano revealed that a 4-session FACT intervention achieved the same clinical outcomes as a 4-session solution-focused brief therapy but had significantly fewer clients drop out of therapy and higher client satisfaction ratings. The PI's previous clinical trial using ACT for Hong Kong parents of children with asthma showed that a 4-session parental training programme using group-based ACT integrated with asthma education was more effective than education alone for improving parental psychological well-being, further proofing the efficacy of a focused and brief ACT intervention. Recently, a feasibility trial (104 participants) of FACT versus waitlist control showed the acceptability and feasibility and provided preliminary data for sample size estimation (see NCT05803252). The present definitive RCT evaluated the effectiveness of Focused ACT versus standard parenting advice.

STUDY AIMS AND HYPOTHESIS TO BE TESTED:

The study's aim is to determine the effectiveness of a video-conferencing Focused Acceptance and Commitment Therapy compared with standard parenting advice for parents of young children with special needs using a robust, randomized controlled trial design.

The hypothesis of the study is that Focused Acceptance and Commitment Therapy (FACT) delivered via videoconferencing will significantly improve parental stress (primary outcome), symptoms of depression, anxiety and psychological flexibility of parents in caring for their children with special needs at multiple intervals: immediately post-intervention, as well as at follow-up assessments six months later, compared to a control group receiving standard parenting advice.

ELIGIBILITY:
Inclusion Criteria:

* Language and Residency: Must be a Cantonese-speaking Hong Kong resident aged 21 years or older.
* Child's age and health status: Must be cohabiting with a preschool or school-aged child (2-9 years old) diagnosed with or suspected of having special needs.
* Caregiver role: Must be the primary caregiver responsible for daily care for the child.
* Technology access: Must have daily access to a smartphone, with either an iPhone or Android operating system, to participate in the study and for potential app-based interventions or communications.

Exclusion Criteria:

* Any parents with severe mental illness, are pregnant, are less than six months postpartum, or have a developmental disability that interferes with their ability to comprehend the programme's content.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Parenting stress | Change from baseline to immediate and 6 months post-intervention
  The Parental Stress Scale (PSS, 18-item, 5-point scale) will be used to assess parenting stress. A higher score represents a higher level of parental stress. The Chinese version of the PSS has demonstrated acceptable psychometric properties and is therefore suitable for use by researchers to assess the parental stress levels of Chinese parents.

SECONDARY OUTCOMES:
Parental depressive symptoms | Change from baseline to immediate and 6 months post-intervention
  The Patient Health Questionnaire (PHQ-9, 9-item, 4-point Likert scale) will be used to assess the frequency of the parents experiencing depressive symptoms in the past two weeks. The Chinese version of the PHQ-9 has demonstrated good internal consistency reliability (Cronbach's alpha = 0.86) and test-retest correlation coefficient (Cronbach's alpha = 0.86).
Parental anxiety symptoms | Change from baseline to immediate and 6 months post-intervention
  The Generalized Anxiety Disorder-7 (GAD-7, 7-item, 4-point Likert scale) will be used to measure the severity of anxiety symptoms. The Chinese version of the GAD-7 demonstrated good reliability and validity with a Cronbach's coefficient of 0.91.
Parental Psychological Flexibility | Change from baseline to immediate and 6 months post-intervention
  The PsyFlex is a 5-point Likert scale with six items to measure the six core processes of Acceptance and Commitment Therapy (ACT): staying present, cognitive defusion, acceptance, self-as-context, values, and committed action. This instrument provides a contextually sensitive measure of psychological flexibility.
ACT Core Process Utilization | Change from baseline to immediate and 6 months post-intervention
  The CompACT-10 is a 10-item, 7-point Likert scale that assesses the critical processes of ACT. This tool has a three-factor structure with internal solid consistency and established convergent and divergent validity with existing measures of ACT processes, as well as indicators of social desirability, psychological distress, and general health and well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong